CLINICAL TRIAL: NCT02258776
Title: Clinical Trial to Determine the Efficacy of Pomegranate for Skin Inflammation and Aging
Brief Title: The Effect of Pomegranate on Aging and Inflammation of the Skin
Acronym: PomSkin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: PomSkin 14-001011
Record Dates: First submitted 2014-09-26; First posted 2014-10-07 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Skin Photoaging, Inflammation and Skin Pathogenic Bacteria
MeSH Terms: conditions — Inflammation | interventions — pomegranate fruit rind

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pomegranate Extract (Active Comparator): 15 healthy subjects, ages 30-45 years who meet all the eligibility criteria in the screening phase of the study will be assigned to the Pomx arm of the study to evaluate the clinical efficacy of pomegranate extract on skin inflammation and aging. Subjects will be asked to take Pomx 1/day for 12 weeks.
  Interventions: Dietary Supplement: Pomegranate Extract
- Pomegranate Juice (Active Comparator): 15 healthy subjects, ages 30-45 years who meet all the eligibility criteria in the screening phase of the study will be assigned to the Pomx arm of the study to evaluate the clinical efficacy of pomegranate juice on skin inflammation and aging. Subjects will be asked to take Pomx 1/day for 12 weeks.
  Interventions: Dietary Supplement: Pomegranate Juice
- Placebo (Placebo Comparator): 15 healthy subjects, ages 30-45 years who meet all the eligibility criteria in the screening phase of the study will be assigned to the Pomx arm of the study to evaluate the clinical efficacy of placebo on skin inflammation and aging. Subjects will be asked to take Pomx 1/day for 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Pomegranate Extract — Pomegranate extract 1000mg will be taken 1/day for 12 weeks.
  Arms: Pomegranate Extract
Dietary Supplement: Pomegranate Juice — Pomegranate juice 8oz will be consumed 1/day for 12 weeks.
  Arms: Pomegranate Juice
Dietary Supplement: Placebo — Placebo will be taken 1/day for 12 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy of pomegranate extract and pomegranate juice on skin inflammation and aging. The information gained from this study may lead to the development of a pomegranate product that can decrease the effects of aging, inflammation and harmful bacteria on the skin.

In this study, two pomegranate products (extract and juice) will be compared with a placebo, a study product that looks like pomegranate extract, but contains no active ingredients.

DETAILED DESCRIPTION:
Pomegranate (Punica granatum L.) is grown commercially in the Near East, India, Spain, Israel and the United States (California) where it is of significant economic importance1. Pomegranate fruits and products, including juice, tea, wine and extracts are widely consumed and recognized for their health benefits. Pomegranate (Punica granatum L.) fruit possesses strong antioxidant, anti-inflammatory and antiproliferative properties. In recent years, most health advantages of pomegranate have been attributed to the presence of ellagitannins, mainly punicalagins and ellagic acid. Punicalagin is unique to pomegranate and is part of a family of ellagitannins. The ellagitannins are hydrolyzed to ellagic acid in the gut, and further metabolized by the colon microflora to form urolith A and B. Investigations using pure bacterial cultures have shown that pomegranate by-products and punicalagins significantly inhibited the growth of pathogenic Escherichia coli, Pseudomonas aeruginosa, clostridia and Staphylococcus aureus.

Oral feeding of pomegranate fruit extract to mice afforded protection to mouse skin against the adverse effects of ultraviolet-B (UVB) radiation by modulating UVB-induced signaling pathways.5 Hydroalcoholic extract based-ointment from pomegranate was reported improving wound healing in vivo. Pomegranate ellagitannins have been demonstrated to have antimicrobial activity. Punicalagin is unique to pomegranate and is part of a family of ellagitannins. The ellagitannins are hydrolyzed to ellagic acid in the gut, and further metabolized by the colon microflora to form urolith A and B. Investigations using pure bacterial cultures have shown that pomegranate by-products and punicalagins significantly inhibited the growth of pathogenic Escherichia coli, Pseudomonas aeruginosa, clostridia and Staphylococcus aureus.

Pomegranate Extract (POMx) is made from pomegranate fruit as a byproduct of pomegranate juice (PJ) production. A second pressing of the fruit liberates a complex mixture of hydrolysable polyphenolic compounds normally ingested with pomegranate juice, and these are purified by spray drying. POMx powder is encapsulated for oral administration, with each capsule containing 1,000 mg of pomegranate polyphenols. The present study will determine whether a pomegranate product (POMx or PJ) can decrease skin photoaging, inflammation and skin pathogenic bacteria.

ELIGIBILITY:
Inclusion Criteria:

1. Age 30-45 years or older, female and any racial/ethnic group
2. Subjects must understand and sign the informed consent prior to participation
3. Subjects must be in generally good health
4. Subjects must be able and willing to comply with the requirements of the protocol.

Exclusion Criteria:

1. Oral or topical retinoid use within twelve months of entry into the study
2. Non-compliant subjects
3. Taking any antibiotics or other medication or dietary supplements regularly
4. Subjects with a significant medical history or concurrent condition that the investigator(s) feel is not safe for the study
5. Subjects who cannot avoid excessive exposure to either natural or artificial sunlight.
6. Allergic to pomegranate products

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2015-10; Primary Completion 2017-02-27 (Actual); Study Completion 2017-02-27 (Actual)

PRIMARY OUTCOMES:
Change in inflammatory markers between pomegranate extract and pomegranate juice versus placebo. | Baseline and 12 weeks
  Utilization of a two-sample t-test to compare the change in between the three groups

SECONDARY OUTCOMES:
Linear mixed effects models to evaluate effect of treatment of time trends and demographic covariates | Baseline and 12 weeks
  Correlation between outcomes measures (e.g. between acne lesion count and skin microbiota) with mixed effects models

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, M.D., Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Center for Human Nutrition, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No